CLINICAL TRIAL: NCT01566968
Title: Novel Endpoints in Cough Challenge Testing.
Acronym: NEAT
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: NEAT Version 2, 18/03/11
Record Dates: First submitted 2012-01-24; First posted 2012-03-30 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Healthy; Chronic Cough; Smokers
Keywords: COPD; Asthma; Healthy volunteers; Chronic cough; Smokers; Cough challenge; Cough challenge testing.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy Volunteers: Adults between ages of 18-75 inclusive who have never smoked and have no history of any respiratory disease for which they are on regular treatment.
  Interventions: Other: Cough challenge test; Other: 24 hour ambulatory cough recording; Other: Cough quality of life questionnaire
- Asthma: Adults between the ages on 18-75 inclusive who have a physician diagnosis of asthma and have no smoking history or minimal smoking history (less than 10 pack years or in other words less than 20 cigarettes per day for 10 years).
  Interventions: Other: Cough challenge test; Other: 24 hour ambulatory cough recording; Other: Cough quality of life questionnaire
- COPD: Adults between the ages of 18-75 inclusive who have previously been smokers (at least 20 pack years) and have physician diagnosis and spirometry evidence of COPD.
  Interventions: Other: Cough challenge test; Other: 24 hour ambulatory cough recording; Other: Cough quality of life questionnaire
- Healthy smokers: Adults between the ages of 18-75 inclusive who are currently smokers (at least 10 pack years history)but have no history of any respiratory disease and no evidence of COPD on spirometry.
  Interventions: Other: Cough challenge test; Other: 24 hour ambulatory cough recording; Other: Cough quality of life questionnaire
- Chronic cough: Adults between ages of 18-75 inclusive who have history of dry cough for at least 8 weeks and have a normal chest x ray and no smoking history or minimal smoking history (less than 10 pack years).
  Interventions: Other: Cough challenge test; Other: 24 hour ambulatory cough recording; Other: Cough quality of life questionnaire

INTERVENTIONS:
Other: Cough challenge test — Cough challenge will be performed with Capsaicin, citric acid and prostaglandin E2.
Other: 24 hour ambulatory cough recording — Cough recording by using an ambulatory sound recording device.
Other: Cough quality of life questionnaire — questionnaire designed to assess impact of cough on a person's life

SUMMARY:
The sensitivity of a person's cough reflex can be measured by getting them to breathe in (inhale) irritant chemicals. There are different methods by which subjects are asked to inhale these chemicals, either by taking one deep breath in, or by asking them to just continue to take a number of breaths. The purpose of this clinical research study is to see if the coughing responses are different in healthy people and people with respiratory problems that make them cough when they are given these chemicals in these two methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 and over.

Meet criteria for subject groups as outlined below:

Healthy volunteers:

* Must be non smokers.
* No history of respiratory disease.

Healthy smokers:

* Current smokers with at least 10 pack year history of smoking.
* Spirometry within normal limits i.e. FEV1 > 80% predicted and FEV1/FVC ratio of > 75% predicted.

Asthma:

* Physician diagnosis of asthma
* Stable asthma.
* Airway hyperresponsiveness to methacoline; PC20< 16mg/ml.
* Non smokers or ex-smokers with smoking history of less than 10 pack years.

COPD:

* Physician diagnosis of COPD
* Ex smokers with smoking history of at least 20 pack years
* Spirometry demonstating evidence of airflow obstruction i.e. FEV1/FVC ratio of < 70%

Chronic cough:

* History of dry cough for at least 8 weeks.
* Normal chest x ray.
* Non smokers or ex smokers of less than 10 pack years history of smoking.

Exclusion Criteria:

* Symptoms of upper respiratory tract infection within the last 4 weeks.
* Participation in another clinical trial of an investigational drug within 4 weeks.
* Use of medication likely to alter cough reflex sensitivity i.e. ACE inhibitors, codeine phosphate, morphine sulphate.
* Patients with severe respiratory disease i.e. FEV1 < 1.0 litre.
* Use of steroid tablets in previous 2 months or taken more than 3 courses of steroid tablets in the preceding 12 months in subjects with asthma or COPD.
* Change in asthma treatment in the preceding 6 weeks in asthma group
* Significant medical co-morbidities likely to affect ability to participate in the trial or affect cough reflex sensitivity e.g. diabetes, stroke, Parkinson's disease, multiple sclerosis etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected from secondary care.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saifudin Khalid, MRCP, Principal Investigator — University Hospital of South Manchester; Ashley Woodcock, MD, Study Chair — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Greater Manchester, United Kingdom